CLINICAL TRIAL: NCT00963638
Title: Beneficial Effects of Magnesium Supplementation On Idiopathic Muscle Cramps
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Corewell Health East (Other)
Responsible Party: Principal Investigator, Rosenbaum, Lewis MD, Principal Investigator, Corewell Health East
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HIC #2008-287
Record Dates: First submitted 2009-08-18; First posted 2009-08-21 (Estimated); Results first posted 2011-06-13 (Estimated); Last update posted 2012-10-01 (Estimated); Status verified 2012-09

CONDITIONS: Muscle Cramp
MeSH Terms: conditions — Muscle Cramp

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- MagTabSR (Experimental)
  Interventions: Dietary Supplement: MagTabSR
- Sugar Pill (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: MagTabSR — MagTabSR/placebo 168 mgs BID for 6 six weeks
  Arms: MagTabSR
Dietary Supplement: Placebo — MagTabSR/placebo 168 mgs BID for 6 six weeks
  Arms: Sugar Pill

SUMMARY:
The goal of this study is to evaluate the effectiveness of magnesium supplements (MagTabSR 168 mgs twice daily) for relief and/or improvement in the frequency, duration, and intensity of chronic leg cramps. Improvement in sleep disturbances and quality of life will also be evaluated.

DETAILED DESCRIPTION:
Chronic leg cramps are prevalent among the aging population affecting sleep patterns and quality of life. Magnesium deficiency may cause muscle weakness and cramps. Magnesium supplementation will be evaluated for the relief and/or improvement of symptoms. The primary objective is to evaluate the efficacy of magnesium supplementation, MagTabSR, 168mg's twice a day, for the relief and/or improvement in the frequency, duration, intensity of leg cramps. Secondary objectives are to evaluate the improvement in sleep disturbances and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* 40-85 Years Old
* No Kidney Impairment
* 2 or more leg cramps per week for last 30 days

Exclusion Criteria:

* < 40 or > 85 Years Old
* Kidney Impairment
* < 2 leg cramps per week for last 30 days
* Enrolled in another research study
* History of seizure disorder
* Current treatment with Lithium
* Malabsorption or major intestinal disorders
* Significantly elevated magnesium level
* History of allergy to magnesium compound
* Use of Quinine for leg cramps
* History of significant diarrhea
* History of drug or alcohol abuse in the last 2 years
* Currently diagnosed with a terminal illness

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-04; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lewis Rosenbaum, MD, Principal Investigator — Physician

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment took place in a private practice clinic between April 15, 2009, and October 5, 2009. Potential study patients responded to a radio advertisement for the study.
Pre-assignment Details: Patients consented were asked to keep a daily diary for 1 week which documented frequency, duration, and severity of leg cramps. Blood was also drawn during this visit to assure values within range. At the second visit, patients who were within range for labs and meet the frequency/duration/severity of leg cramps were randomized.
Groups:
- Magnesium Tablet SR (MagTabSR): MagTabSR is 168mg taken 2 times per day for 30 days
- Sugar Pill: Sugar pill is taken 2 times per day for 30 days
Period: Overall Study
Arm/Group | Magnesium Tablet SR (MagTabSR) | Sugar Pill
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Magnesium Tablet SR (MagTabSR) | Sugar Pill | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 7 | 14
  >=65 years | 13 | 13 | 26
Age Continuous [Mean (Standard Deviation); unit: years] | 67.25 (9.9) | 66.00 (9.3) | 66.62 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 13 | 23
  Male | 10 | 7 | 17
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Change in Frequency of Leg Cramps
Description: Patients recorded number of leg cramps daily. The primary outcome measure was changed to the weekly average number of daily leg cramps for the first 28 days (4 weeks) after the start of treatment compared to the week prior to treatment (week 4 - pretreatment baseline).
Time Frame: 30 days
Measure: Mean (Standard Deviation); unit: Cramps per week
Arm/Group | Magnesium Tablet SR (MagTabSR) | Sugar Pill
Number analyzed (Participants) | 20 | 20
Cramps per week | .99 (1.13) | .53 (.52)

2. Primary Outcome: Frequency/Duration of Muscle Cramps
Time Frame: 30 days
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Magnesium Tablet SR (MagTabSR) | Sugar Pill
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No